CLINICAL TRIAL: NCT00516152
Title: Phase II Study Evaluating Busulfan and Fludarabine as Preparative Therapy in Adults With Hematopoietic Disorders Undergoing Matched Unrelated Donor Stem Cell Transplantation
Brief Title: Phase II Study Evaluating Busulfan and Fludarabine as Preparative Therapy in Adults With Hematopoietic Disorders Undergoing MUD SCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Beth Davis, University of California San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-2214
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2009-01-26 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Myeloid Leukemia; Acute Myelogenous Leukemia; Myelodysplasia; Acute Lymphocytic Leukemia; Severe Aplastic Anemia; Non-Hodgkin's Lymphoma; Lymphoproliferative Disease; Multiple Myeloma; Advanced Myeloproliferative Disease
Keywords: Matched Unrelated Donor; Stem Cell Transplantation; Busulfan; fludarabine; Hematopoietic Disorder
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Aplastic; Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Multiple Myeloma | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Busulfan/Fludarabine phosphate/Tacrolimus/Methotrexate/G-CSF — Day Preparative Regimen for GVHD Prophylaxis
  * 7 Busulfan 0.8 mg/kg IV Q6 hurs, Fludarabine 30 mg/m(2)IV
  * 6 Busulfan 0.8 mg/kg IV Q6 hurs, Fludarabine 30 mg/m(2)IV
  * 5 Busulfan 0.8 mg/kg IV Q6 hurs, Fludarabine 30 mg/m(2)IV
  * 4 Busulfan 0.8 mg/kg IV Q6 hurs, Fludarabine 30 mg/m(2)IV
  * 3 Fludarabine 30 mg/m(2)IV
  * 2 REST Tacrolimus 0.01 mg/kg CIVI
  * 1 REST 0 Unrelated Stem Cell/Bone Marrow Infusion
    * 1 Methotrexate 5mg/m(2)IV
    * 3 Methotrexate 5mg/m(2)IV
    * 6 Methotrexate 5mg/m(2)IV
    * 7 G-CSF 5mcg/kg SQ daily
    * 11 Methotrexate 5mg/m(2)IV
    * 90 Evaluate Response

SUMMARY:
The primary objective of this study is to assess the safety and efficacy of performing unrelated stem cell transplants using intravenous busulfan and fludarabine as preparative therapy and tacrolimus plus methotrexate as the GVHD prophylaxis regimen. The goal is to demonstrate safety, aiming for a transplant related mortality rate (TRM) of < or equal to 40% at 100 days. A TRM of > or equal to 60% will be considered unacceptable. Another goal is to demonstrate efficacy by showing and overall survival of >40% at 1-year following transplant.

ELIGIBILITY:
Inclusion Criteria:

* No fully or single-antigen mismatched sibling donor is available to donate stem cells.
* Age >15 and <61
* ECOG PS < or equal to 2
* Adequate renal function with serum creatinine <2.0 mg/dl
* Pulmonary diffusing capacity >40% of predicted
* Cardiac ejection fraction >40% as measured by radionuclide wall motion study or echocardiography
* No active liver disease. Total bilirubin must be < or equal to 2.0 mg/dl. Alkaline phosphatase and AST must be less than three times the upper limit of normal. Patients with hepatitis C and active hepatitis B are eligible only if a liver biopsy is performed and there is < or equal to grade 2 inflammation. Patients wtih a history of HBV infection should be tested for HBeAg, antiHBe and HBV DNA (quantitative). Patients with active HBV viral replication should receive anti-viral therapy.
* Negative serology for the human immunodeficiency virus (HIV)
* Available HLA-matched donor (see HLA compatibility requirements below)
* Signed informed consent from the recipient

Exclusion Criteria:

* Ongoing active infection
* Pregnancy and/or nursing
* Active, uncontrolled CNS leukemia
* Opinion of BMT Committee that autologous or mini-allogeneic transplant would be the preferable form of treatment
* Receipt of any chemotherapy within 3 weeks of study entry except for hydroxyurea or imatinib mesylate. Use of interferon within 3 months of starting therapy.

Ages: 15 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2002-11; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G. Martin, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- See also: UCSF Cancer Center Home Page — http://cancer.ucsf.edu